CLINICAL TRIAL: NCT01353638
Title: An Open Label, Randomized, Two-Period Crossover Study to Evaluate the Safety and Efficacy of the Addition of Alanyl-Glutamine-Dipeptide to Dialysis Solutions in Peritoneal Dialysis (PD) (Ala-Gln in PD)
Brief Title: Safety and Efficacy of the Addition of Alanyl-Glutamine-Dipeptide to Dialysis Solution in Peritoneal Dialysis
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Primary endpoint (HSP) could not be analyzed with the specified method in the planned interim analysis; a method of increased sensitivity had to be established.
Sponsor: Christoph Aufricht (Other)
Responsible Party: Sponsor-Investigator, Christoph Aufricht, Ao.Univ.-Prof. Dr.med.univ., Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Ala-Gln in PD
Record Dates: First submitted 2011-05-05; First posted 2011-05-13 (Estimated); Last update posted 2015-09-11 (Estimated); Status verified 2015-09

CONDITIONS: End Stage Renal Disease
Keywords: Peritoneal dialysis; Alanyl-Glutamine-Dipeptide; Heat shock protein; Peritoneal cells; functional maintenance of the peritoneal membrane
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — alanylglutamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Other): Arm A includes 14 patients. In treatment period 1, arm A receives standard PDF with the interventional drug alanyl-glutamine-dipeptide as add-on. As it is a cross-over study design, in treatment period 2, group A receives standard PDF without add-on.
  Interventions: Drug: Dipeptiven (Alanyl-glutamine-dipeptide)
- Arm B (Other): Arm B includes 14 patients who in treatment period 1 receive standard PDF without the investigational drug. As it is a cross-over study design, in treatment period 2 arm B receives standard PDF with alanyl-glutamine-dipeptide as add-on.
  Interventions: Drug: Dipeptiven (Alanyl-glutamine-dipeptide)

INTERVENTIONS:
Drug: Dipeptiven (Alanyl-glutamine-dipeptide) — Two arms (A and B) and two treatment periods (1 and 2) are scheduled for this study. Each arm includes 14 patients. Schedule arm A: Treatment period 1 with one single peritoneal dialysis exchange (standard PD solution) with Alanyl-Glutamine-Dipeptide as add-on. 17,4 ml Dipeptiven (=3,48g N(2)-L Alanyl-L-Glutamin) will be dissolved at a final concentration of 0,174 %(= 8 mmol/l) in 2 liters of Dianeal®PD4 (at PH:5,5; Glucose-Concentration 3,86 %). After a wash out period (28 days + max 7 days), arm A undergoes treatment period 2, that is one single peritoneal dialysis exchange with standard PD solution without Alanyl-Glutamine-Dipeptide. Schedule Arm B: Treatment period 1 with one single peritoneal dialysis exchange with standard PD solution without Alanyl-Glutamine-Dipeptide followed by wash-out. Treatment period 2 for arm B includes one single peritoneal dialysis exchange with standard PD solution with Alanyl-Glutamine-Dipeptide as add-on. Dosages remain exactly the same.
  Other Names: Standard PD solution: Dianeal® PD4 Glukose 3,86%

SUMMARY:
Peritoneal dialysis (PD) is a cost effective and safe form of renal replacement therapy in patients suffering from end stage renal disease.

However currently available PDF (peritoneal dialysis fluids) are not biocompatible for the peritoneal cavity and its cells. Acute cytotoxic effects of the majority of the current glucose-based PDF are caused by low pH, lactate, high glucose and its degradation products (GDP).

Toxic effects of PDF can thus be extended to suppression of mesothelial HSR (heat shock reactions) following PDF exposure resulting in increased susceptibility of mesothelial cells against PDF exposure: PDF inherent stress factors fail to adequately induce HSP as effectors of the cellular stress response - the adequate HRS rather seems to be blocked.

Hence, therapeutic approaches to activate and enhance the HSR will reduce peritoneal damage and organ failure and improve the survival of organisms.

Preclinical results demonstrated that supplementation of PDF with pharmacological doses of alanyl-glutamine restored HSP expression and increased the resistance of mesothelial cells in in-vitro models of PD and preserved peritoneal integrity in in-vivo models of PD.

After these positive preclinical results, this study shall now clarify, whether the addition of alanyl-glutamine to the most commonly used glucose-based PDF is safe and tolerable. Therefore PDFs will be drained in a randomized cross-over study. Main outcomes measures will be total HSP expression in peritoneal cells and changes of the peritoneal transport kinetics and the presence/absence/severity of side effects.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to any study-mandated procedure
* Male and female patients aged ≥ 19 years old
* Chronic renal failure; 2 months stable on PD
* no peritonitis within the previous 2 months
* Without severe concomitant disease
* Negative pregnancy test in female patients of childbearing potential and adequate contraception in female patients of childbearing age

Exclusion Criteria:

* Known hypersensitivity to study medication
* Treatment with another investigational drug within 1 month prior to start of study medication
* Malignancy requiring chemotherapy or radiation
* Pregnancy or nursing,
* Presumed non-compliance
* Limited efficacy of peritoneal dialysis due to anatomical anomalies or severe intra-abdominal adhesions
* Clinical significant inflammatory parameters
* Less than 50 kg body weight
* Immunosuppressive therapy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-04; Primary Completion 2012-03 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Primary Endpoint: Total heat shock expression in peritoneal cells from dialysate samples; | up to 70 days
  In this study, an increase of total heat shock protein expression will be detected in cells from the peritoneal effluent at 240 min by staining of the cytospin and by Western blot analysis of the cellular pellet of the effluent. Total heat shock expression from dialysate samples is calculated in percent.

SECONDARY OUTCOMES:
Clinical PET-test to measure specific transport kinetics in peritoneal cells (creatinine, urea, sodium, potassium, phosphor, glucose, protein) | up to 70 days
  The ratio of solute concentrations in dialysate and plasma (D/P ratio) at specific times (t) during the dwell signifies the extent of solute equilibration. Creatinine, glucose, urea, electrolytes, phosphate, and proteins are the commonly tested solutes for clinical use, in this study alanine, glutamine and alanyl-glutamine-dipeptide also will be measured to allow assessment of the respective resorption kinetics.
Cell number in peritoneal effluent; | up to 70 days
  At the end of PD, total peritoneal cell count of the dialysate is measured; Unit of measurement: cells/µl
cytokines (IL-6, IL-8, TNFα); | up to 70 days
  At the end of PD cytokines contained in the dialysate are being analysed. Unit of measurement: pg/ml
Cell function (phagocytosis and cytokine production) | up to 70 days
  Analysis of cell function in dialysate at the end of PD by declaring the contingent of positive cell function in percent;
Morphology of peritoneal cells from effluent (cell culture) | up to 70 days
  At the end of PD, the cells contained in the dialysate are being differentiated in following categories: ephitelium; non epithelium; mixed.
Biomarker CA125 | up to 70 days
  At the end of PD, the amount of CA125 in the dialysate is measured in U/ml.
Tolerability/safety endpoints: No. and severity of AEs | up to 70 days
  During the trial and after signing informed consent, the presence/absence/severity of AEs occurring to patients is being documented. Measurement parameter is no. and severity of AEs (including SAEs and SUSARs).

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Aufricht, Univ.Prof.Dr., Study Director — Medical University of Vienna
Locations (1):
- Department of Internal Medicine III; Clinical Division of Nephrology and Dialysis; Medical University of Vienna, Vienna, Austria

REFERENCES:
- See also: Related Info — http://www.meduniwien.ac.at